CLINICAL TRIAL: NCT03868566
Title: An Open-Label Study to Assess the Hepatic Protection Effect of a Food Supplement Product, SNP-612, in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: An Open-Label Study to Assess the Hepatic Protection Effect of SNP-612, in Patients With NAFLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment difficulties due to Covid-19
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNP-612-202
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Experimental: SNP-612 dose1 Experimental: SNP-612 dose2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SNP-612 dose1 (Experimental): dose1 once a day orally for 12 weeks
  Interventions: Drug: SNP-612 dose1
- SNP-612 dose2 (Experimental): dose2 once a day orally for 12 weeks
  Interventions: Drug: SNP-612 dose2

INTERVENTIONS:
Drug: SNP-612 dose1 — Subjects will take dose1 once a day orally for 12 weeks
  Arms: SNP-612 dose1
Drug: SNP-612 dose2 — Subjects will take dose2 once a day orally for 12 weeks
  Arms: SNP-612 dose2

SUMMARY:
The primary objective of the study is to compare the changes in ALT to baseline among patients with non-alcoholic fatty liver disease (NAFLD) following the 3-month treatment of 3 different dosing regimens of SNP-612. The secondary objectives will be to compare the changes in other liver function tests, cytokeratin-18 (CK-18) fragment level and adverse event / serious adverse event rates.

DETAILED DESCRIPTION:
An open-label study will be conducted in medical centers around Taiwan. The objective of the study is to investigate the efficacy and safety of SNP-612 for the treatment of NAFLD.

Subjects who fulfill all the entry criteria and have written informed consent will be enrolled to the study. Considering a 10% drop-out rate, approximately 72 subjects will be enrolled in order to recruit 64 evaluable subject subjects to complete the enrollment.

Subjects will be administered the study agents oral daily for 3 months or until treatment terminates prematurely. Subjects will return to the study center for clinical evaluation once every 4 weeks throughout the treatment period. Clinical assessment procedures and laboratory tests including ultrasound imaging, hematology with differential, biochemistry, liver function panel, and urinalysis, will be performed at each study visit. The primary endpoint assessment will be the reduction of ALT, at completion of Week 12 compared to baseline. With 64 evaluable patients, there will be an 80% chance of detecting a significant difference at a two sided 0.05 significance level.

Subjects who finish treatment or discontinue prematurely from the study for any reason after receiving one or more doses of study agent will be assessed for safety for 2 (±1) weeks after the last study agent dose or longer in the case of any significant AE or abnormal biochemical or clinical finding.

Each subject will participate in the study for approximately 14 weeks (including the enrollment/baseline visit, 3 routine monthly visits during treatment period, and 1 follow-up visit after 2 weeks of the end of treatment).

It is assumed the study will include a 6 months enrollment period and a further 4 months to complete the follow-up for all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Body weight ≥ 54 kg
3. Diagnosis of non-alcoholic steatohepatitis (NASH) as evidenced by imaging or other diagnostic assessments. Subject should have documented liver fat content ≥ 10.0 % as measured by MRI method prior to study agentagent administration.
4. Phenotypic diagnosis of NASH based on one or more of the following:

   1. Alanine aminotransferase (ALT) levels ≥ 1.5x upper limit of normal (ULN) on at least two occasions, seven or more days apart, prior to study agent administration
   2. ALT ≥ ULN on at least two occasions, seven or more days apart, prior to study agent administration AND body mass index (BMI) ≥ 25 AND diagnosis of Type 2 DM
5. Have adequate organ functions as defined by the following examinations prior to the start of study treatment:

   1. Hematology: Hemoglobin ≥ 9 g/dL, a platelet count ≥ 100 x 10^9/L, and a white blood cell count ≥ 3.0 x 10^9/L
   2. Renal: creatinine clearance ≥ 90 mL/min (by Cockcroft-Gault equation), serum uric acid < 9.0 mg/dL
6. Able to provide written informed consent, and understand and comply with the requirements of the study

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to enter the study:

1. Decompensated or severe liver disease as evidenced by one or more of the following:

   1. Confirmed cirrhosis or suspicion of cirrhosis
   2. Liver transplant
   3. Liver malignancy
   4. Ascites
   5. Bilirubin > ULN, or ALT or AST > 5 x ULN, or Alkaline phosphatase (ALP) > 2x ULN
   6. Acute or chronic hepatitis A, B, C, HIV, or other liver diseases affecting liver function.

   Patients with cysts, hemangiomas, or similar abnormalities, are accepted.
2. History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120-mL wine or 14 cans of 350-mL beer), or other substance abuse within the prior two years
3. Subjects who are unable to undergo an MRI scan.
4. Subjects have electronically, magnetically and mechanically activated implanted devices, including but not limited to automatic cardioverter defibrillators, cardiac pacemakers, insulin pumps, metallic splinters in the eye, ferromagnetic haemostatic clips in central nervous systems or vascular vessels.
5. Significant systemic or major illness other than liver disease, including auto-immune disease, coronary artery disease, cerebrovascular disease, malignant neoplasms, pulmonary disease, renal insufficiency, serious psychiatric disease, and/or other serious disease, that, in the opinion of the Investigator would preclude the subject from participating in and completing the study
6. Documented history of serious allergic reaction to SNP-612 or any structurally related compounds
7. Diabetic patients who have not maintained a stable dose of oral medication for hyperglycemia or have had more than 10 percent change in their insulin dose over the past two months
8. Regular use of agents that are potent against hepatitis or affecting lipid metabolisms, including but not limited to HMGCoA reductase inhibitors (statins), fibrates, silymarin, N-acetylcysteine, or anti-TNF therapies.
9. Pregnant or lactating
10. Female of child-bearing potential who are not committed to taking reliable contraception during the participation of the study and at least 4 weeks after the end of the study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Change in serum ALT | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition

SECONDARY OUTCOMES:
Change in serum AST | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition
Change in serum Alk-P | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition
Change in serum γ-GT | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition
Change in GSP | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition
Change in liver fat content as measured by liver fat fraction (FF) with magnetic resonance imaging method. | 12 weeks
  A non-invasive method will be utilized to estimate liver fat content (%) by MRI calculated liver FF.
Change in serum CK-18 fragment levels | 12 weeks
  A reduction from baseline (i.e. a negative percent value) indicates an improvement in condition
Rate of AE/SAE | 12 weeks
  Rate of patients who experience AE/SAE at end of treatment
Rate of AEs leading to discontinuation at end of treatment | 12 weeks
  Rate of patients who experience AEs leading to discontinuation at end of treatment

OTHER OUTCOMES:
Insulin resistance | 12 weeks
  Change in insulin resistance at Week 12
Triglycerides | 12 weeks
  Change in serum at Week 12
Low density lipoprotein | 12 weeks
  Change in serum at Week 12
Total cholesterol | 12 weeks
  Change in serum at Week 12
High density lipoprotein | 12 weeks
  Change in serum at Week 12
Gene expression biomarkers | 12 weeks
  Gene expression biomarkers (ACC1, Adfp, AOX, Cat, CCL20, CCR2, Cpt1α, CYP2E1, CYP4A11, CYP7A, Dgat1, Dgat2, FAS, Gapdh, Gpx1, Gpx2, Gpx3, Gpx4, GSS, Hadh, Ho1, HSL, IL-10, IL-1β, IL-6, iNOS, LCAD, NF-κB1, NF-κB2, Pparα, PPARβ/δ, PPARγ, SCD-1, Sod1, Sod2, Sod3, SREBP-1c, TGFβ, TLR4, TNFα, Ucp2, VLCAD, α-SMA, β-actin) related to NASH changes in blood at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Lueng Shih, MD,PhD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho HT, Shih YL, Huang TY, Fang WH, Liu CH, Lin JC, Hsiang CW, Chu KM, Hsiong CH, Chen GJ, Wu YE, Hao JY, Liang CW, Hu OY. Mixed active metabolites of the SNP-6 series of novel compounds mitigate metabolic dysfunction-associated steatohepatitis and fibrosis: promising results from pre-clinical and clinical trials. J Transl Med. 2024 Oct 14;22(1):936. doi: 10.1186/s12967-024-05686-7. PMID 39402603